CLINICAL TRIAL: NCT01998295
Title: Parasite Clearance Time and Time to Recurrent Infection Following Treatment With Artemether/Lumefantrine Among Children With Uncomplicated P. Falciparum Malaria Five Years After Wide Scale Use of the Drug in Tanzania
Brief Title: Parasite Clearance Time and Time to Recurrent Infection Following Treatment With Artemether/Lumefantrine
Acronym: PCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Richard Mwaiswelo, Investigator, Muhimbili University of Health and Allied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.0.2011
Record Dates: First submitted 2013-11-15; First posted 2013-11-28 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Instantaneous Clearance
Keywords: Clearance time; Recurrence time; Artemether/lumefantrine; P. falciparum; Uncomplicated malaria; Children
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artemether/lumefantrine (Active Comparator): Artemether/lumefantrine tablets, 6 doses, for 3 days
  Dosage:
  1. tablet for body weight between 5-14.9 Kilograms.
  2. tablets for body weight between 15-24.9 Kilograms.
  3. tablets for body weight between 25-34.9 Kilograms.
  Interventions: Drug: Artemether/lumefantrine

INTERVENTIONS:
Drug: Artemether/lumefantrine — Medication was given at 0, 8, 24, 36, 48 and 60 hours. Food was given to all patients prior to medication to ensure proper absorption of the drug.
  Other Names: Coartem

SUMMARY:
Plasmodium falciparum resistance against artemisinins has been confirmed in South-East Asia and it is expressed phenotypically as a slow rate of parasite clearance. Nonetheless, it is not known whether the problem exist in Tanzania. This study assessed parasite clearance time and time to recurrent infection following treatment with Artemether/Lumefantrine (AL) among children with uncomplicated malaria.

DETAILED DESCRIPTION:
Artemether/Lumefantrine (AL) has been in wide scale use in Tanzania since 2007 as first line treatment for uncomplicated falciparum malaria. Nonetheless, reports of confirmed resistance against Artemisinin derivatives expressed phenotypically as prolonged parasite clearance have emerged from South-East Asia (SEA), signifying reduced parasites susceptibility to the otherwise rapidly acting artemisinins. Prolonged clearance is associated with an increase in day 28 treatment failure, gametocytes carriage and transmission of resistance. Nonetheless, no detailed study has been done in East Africa to assess parasite clearance time following treatment with Artemisinin based combination therapies (ACTs).

In order to evaluate time to parasite clearance following treatment with AL, we conducted a detailed clinical trial with twenty blood sampling time points prior, during and after treatment. Detailed sampling allowed us to assess parasite clearance, and selection of Plasmodium falciparum multidrug resistance (Pfmdr) 1 N86Y and Plasmodium falciparum chloroquine resistance transporter (Pfcrt) K76T genes between different time points and its association with parasite clearance and recurrence. Furthermore, as a sensitive tool and an ideal early warning system, nested polymerase chain reaction (PCR) was used to assess parasite clearance and compare it with microscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-120 months
* Presence of asexual P. falciparum parasitaemia of 2000-200 000/μL
* No general danger signs or severe malaria present
* Hemoglobin ≥5 g/dL
* History of fever within 24 hours or axillary temperature ≥ 37.5 degree Celsius
* No other cause of fever is detectable
* No severe malnutrition
* Guardian/patient has consented

Exclusion Criteria:

* general danger signs or signs of severe falciparum malaria
* severe malnutrition
* febrile condition due to diseases other than malaria
* regular medication which might interfere with antimalarial pharmacokinetics
* contraindications to any medicine being used

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time to parasite clearance | 72 hours
  Time to parasite clearance was assessed by taking blood samples and examining it by light microscopy prior (0 hour) and during treatment at 4, 8, 12 hours and then 6 hourly until two consecutive negative blood slides.

SECONDARY OUTCOMES:
Time to recurrent infection | 42 days
  Time taken for parasites to reappear in the peripheral blood of the participant after initial treatment was assessed during the 42 days of follow up from blood samples taken on days 14, 21, 28 and 42.

OTHER OUTCOMES:
Time to parasite clearance | 7 days
  Blood samples collect on filter papers prior (0 Hour), during and after medication at 4, 8, 12 and after every 6 hours until 72 hours and on day 7 were analyzed by PCR to assess parasite clearance. Parasite positivity after day 7 was considered as recurrent infection.
Time to alleles clearance | 168 hours
  Time to clearance of parasites carrying Pfmdr 1 N86Y and Pfcrt K76T alleles was assessed by molecular genotyping using blood samples collected during the early phase of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Martensson, PhD, Study Director — Karolinska Institutet
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Mwaiswelo R, Ngasala B, Jovel I, Xu W, Larsson E, Malmberg M, Gil JP, Premji Z, Mmbando BP, Martensson A. Prevalence of and Risk Factors Associated with Polymerase Chain Reaction-Determined Plasmodium falciparum Positivity on Day 3 after Initiation of Artemether-Lumefantrine Treatment for Uncomplicated Malaria in Bagamoyo District, Tanzania. Am J Trop Med Hyg. 2019 May;100(5):1179-1186. doi: 10.4269/ajtmh.18-0729. PMID 30860013